CLINICAL TRIAL: NCT00239408
Title: Spiriva Assessment of FEV1 - (SAFE-Portugal). The Effect of Inhaled Tiotropium Bromide (18 Mcg Once Daily) on the Change in FEV1 During Treatment in Patients With COPD. A Three-month Parallel Group, Double-blind, Randomised, Placebo-controlled Study.
Brief Title: Spiriva (Tiotropium Bromide) Assessment of FEV1 - (SAFE-Portugal).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.282
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Function Tests; Tiotropium Bromide

INTERVENTIONS:
Device: Pulmonary function Testing
Drug: tiotropium bromide

SUMMARY:
Evaluate whether the effect of inhaled tiotropium bromide on the change in trough forced expiratory volume (FEV1), compared to placebo in patients with chronic obstructive pulmonary disease (COPD), is affected by smoking status.

DETAILED DESCRIPTION:
Evaluate whether the effect of inhaled tiotropium bromide on the change in trough FEV1 from baseline to week 12 compared to placebo in patients with COPD is affected by smoking status. Secondary objectives include FEV1 at interim visit and FVC at on-treatment visits, use of rescue medication, COPD symptom scores, Physicians Global Evaluation and EQ-5D scores.

Study Hypothesis:

The primary objective of the study is to show superiority of tiotropium against placebo with respect to trough FEV1 at 12 weeks. Then the 5% two-sided hypotheses test is:

H0: Mean trough FEV1 at 12 weeks in tiotropium = Mean trough FEV1 at 12 weeks in placebo H1: Mean trough FEV1 at 12 weeks in tiotropium unequal Mean trough FEV1 at 12 weeks in placebo If the null hypothesis is rejected in favour of the alternative hypothesis (H1) based on all patients, the same hypotheses will be tested in both sub-populations of current and ex-smokers respectively.

Comparison(s):

Tiotropium bromide - 18 mcg capsule inhaled via the HandiHaler vs Placebo powder capsules for oral inhalation, via the HandiHaler.

ELIGIBILITY:
Main Inclusion criteria: 1.Diagnosis of chronic obstructive pulmonary disease. 2.Patient is male or female, age <=than 40 years. 3. Patient has a smoking history of <=10 pack-year.4.Patient is able to be trained in the proper use of HandiHaler 5.Patient is able to be trained to perform technically satisfactory spirometry and must be able to maintain records during the study period as required by the protocol. 6.Patient must be willing and able to sign informed consent prior to participation in the study i.e. prior to washout of their usual pulmonary medications.

Main exclusion criteria 1.History of asthma, allergic rhinitis or atopy. 2. A lower respiratory tract infection or any COPD exacerbation in the past 4 weeks prior to Visit 1 or during the two week Screening Period 3.History of life threatening bronchial obstruction, cystic fibrosis or bronchiectasis 4. Oral corticosteroid medication if initiated or modified within the last 6 weeks prior to Visit 1 or if daily dose > 10 mg prednisone or 20 mg or more every other day (or equivalent). 5.Patients who have started or stopped an exercise rehabilitation program within 4 weeks of visit 6.Patients who regularly use daytime oxygen therapy for more than one hour per day and who, in the investigator's opinion, will be unable to abstain from the use of oxygen therapy during testing. 7. Patients who have undergone thoracotomy with pulmonary resection or lobectomy (lung volume reduction surgery). 8.Tuberculosis with indication for treatment. 9. Recent history (i.e. 6 months or less) of myocardial infarction.10. Patients with known moderate or severe renal insufficiency.11. Patients with symptomatic prostatic hypertrophy or bladder neck obstruction. 12.Patients with known narrow-angle glaucoma.13.History of unstable arrhythmia with a life threatening event or change of therapy during the past year.14. History of cancer, other than treated basal cell carcinoma, within the last 5 years 15.Intolerance to anticholinergic containing products, and/or to lactose or any other components of the inhalation capsule delivery system.16.Patients who are being treated with beta-blockers including eye drops.17.Patients who are being treated with antihistamines (H1 receptor antagonists), for asthma or excluded allergic conditions (See Exclusion Criteria No.2).18.Patients who are being treated with monoamine oxidase inhibitors or tricyclic antidepressants.19. Patients who are being treated with oral beta-adrenergics.20. Patients who have taken cromolyn sodium or nedocromil sodium within 1 month of Visit 1.21.Patients who have taken antileukotrienes or leukotriene receptor antagonists within 1 month of Visit 1. 22.Concomitant or recent (within the last month or 6 half lives, whichever is greater) use of investigational drugs prior to the screening visit (Visit 1). 23. Significant alcohol or drug abuse within the past 12 months. 24. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception.24. Previous participation in this study (i.e. randomized).26. Patients who have taken commercially available Spiriva. 27.History of any clinically significant disease, defined as a disease which in the opinion of the investigator may the patient at risk because of participation in the study OR a disease which may influence the results of the study OR the patient's ability to participate in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311
Dates: Start 2002-12; Primary Completion 2004-04 (Actual); Study Completion 2004-04

PRIMARY OUTCOMES:
Change in trough FEV1 after 12 weeks of treatment. | week 12

SECONDARY OUTCOMES:
Trough FEV1 at interim visit | week 6
Change in FVC at weeks 6 and 12 | week 6, week 12
Use of rescue medication (daytime and night-time) | 12 weeks
Assessment of COPD symptoms | week 0, week 6, week 12
The Physician's Global Evaluation at Visits 2 and 4 | week 0, week 12
Quality of life questionnaire (EQ-5D) at Visits 2 and 4 | week 0, week 12
Pulse Rate | 12 weeks
Blood Pressure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Portugal Lda
Locations (33):
- Portugal (33):
  - Hospital Garcia de Orta, Almada
  - Hospital Fernando Fonseca, Amadora
  - Hospital Santo Espírito de Angra do Heroismo, Angra Do Heroismo - Açores
  - Hospital Infante D. Pedro, Aveiro
  - Unidade Funcional de Infecciologia, Barreiro
  - Hospital de S. Marcos, Braga
  - Hospitais da Universidade de Coimbra, Coimbra
  - Centro Hospitalar de Coimbra, Coimbra
  - Centro Hospitalar da Cova da Beira, Covilha
  - Hospital Espírito Santo, Evora
  - Hospital Distrital de Faro, Faro
  - Hospital Distrital da Figueira da Foz, Figueira da Foz Municipality
  - Centro Hospitalar do Funchal, Funchal
  - Hospital de Sousa Martins, Guarda
  - Hospital Senhora da Oliveira, Guimarães
  - Hospital Particular de Lisboa, Lisbon
  - Instituto Português de Oncologia Francisco Gentil, Lisbon
  - Hospital de Santa Marta - HCL, Lisbon
  - Hospital Egas Moniz, Lisbon
  - Hospital Santa Maria, Lisbon
  - Hospital Pulido Valente, Lisbon
  - Unidade Local de Saúde de Matosinhos, Matosinhos Municipality
  - Hospital Divino Espírito Santo, Ponta Delgada - Açores
  - Hospital Barlavento Algarvio, Portimão
  - Hospital Geral de Santo António, Porto
  - Hospital de São João, Porto
  - Hospital Joaquim Urbano, Porto
  - Hospital de S. Sebastião, Santa Maria da Feira
  - Hospital Distrital de Santarém, Santarém
  - Hospital de S. Bernardo, Setúbal
  - Hospital Rainha Santa Isabel, Torres Novas
  - Centro Hospitalar de V. N. de Gaia, V.N.Gaia
  - Hospital de S. Teotónio, Viseu